CLINICAL TRIAL: NCT07224438
Title: Kisspeptin Administration Subcutaneously to Patients With Hypothalamic Amenorrhea
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 565178; R37HD043341 (NIH)
Record Dates: First submitted 2025-11-03; First posted 2025-11-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hypothalamic Amenorrhea; Hypogonadotropic Hypogonadism
Keywords: hypothalamic amenorrhea; hypogonadotropic hypogonadism; kisspeptin
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Kisspeptin pump (Experimental): SC administration of kisspeptin for two weeks (pulsatile)
  Interventions: Drug: kisspeptin 112-121

INTERVENTIONS:
Drug: kisspeptin 112-121 — SC administration of kisspeptin for two weeks (pulsatile, approximately every 90 minutes)
  Other Names: Metastin 45-54

SUMMARY:
The goal of this study is to see whether kisspeptin, a naturally occurring hormone, can stimulate the release of other reproductive hormones in women with hypothalamic amenorrhea (HA). The investigators are also examining whether kisspeptin can help women release eggs from their ovaries. Kisspeptin will be administered subcutaneously (SC) for two weeks in a pulsatile fashion. Ultrasound monitoring of ovarian follicular growth and frequent blood sampling (every 10 minutes for up to two hours) will be performed to assess the physiologic response to kisspeptin over time.

DETAILED DESCRIPTION:
Assignment: All study subjects will undergo the same interventions.

Delivery of Interventions:

* The subject will undergo a review of their medical history, physical exam, and screening laboratories.
* A pelvic ultrasound will be performed to assess baseline follicular size.
* A pump will be placed to administer pulsatile SC kisspeptin for two weeks.
* During the course of kisspeptin administration, subjects will
* Undergo q10 min blood sampling (approximately 4 sessions, 2 hours each)
* Undergo pelvic ultrasounds (approximately 4 sessions)
* Optional q10 min sampling up to 10 hours may take place before and after the course of kisspeptin

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18-45 years
* Acquired HH (hypothalamic amenorrhea, aka functional hypogonadotropic hypogonadism)
* Normal blood pressure (systolic BP < 140 mm Hg, diastolic < 90 mm Hg)
* Hemoglobin no less than 0.5 g/dL below the lower limit of the reference range for normal women
* Negative serum hCG pregnancy test
* No current or recent use of a medication (including hormonal replacement) that, in the opinion of a study investigator, can modulate the reproductive axis OR willing to complete an appropriate washout for that particular medication and its method of administration
* If applicable, willing to use birth control methods (as approved by a study medical professional) during the entire study and for one month after the last dose of study drug

Exclusion Criteria:

* Any condition (medical, mental, or behavioral) that, in the opinion of a study investigator, would likely interfere with participation in/completion of the protocol
* Excessive alcohol consumption (>10 drinks/week)
* Active use of illicit drugs
* Pregnant
* Trying to become pregnant during protocol participation
* Breast feeding
* History of any of the following: bilateral oophorectomy (ovaries were removed), breast cancer, thromboembolic disease, coronary artery disease, stroke, thrombophilic disorders, or undiagnosed abnormal genital bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Change of luteinizing hormone (LH) pulse amplitude | 2 weeks
  Difference in LH amplitude on the first day of kisspeptin administration vs the last day of kisspeptin administration

OTHER OUTCOMES:
The proportion of participants that achieve development of a mature follicle or show evidence of ovulation | 2 weeks
  Mature follicle achievement is defined as evidence of a follicle with maximum diameter ≥18 mm. Evidence of ovulation is defined as detection of a corpus luteum on ultrasound in combination with elevated progesterone level.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No